CLINICAL TRIAL: NCT05455021
Title: Feasibility Study of the Vessel Restoration System (VRS) for the Treatment of Atherosclerotic Lesions in the Superficial Femoral Artery (SFA) and/or Popliteal Artery (PA) After Sub-optimal Percutaneous Transluminal Angioplasty (PTA) or Atherectomy: REACTIVATE I
Acronym: REACTIVATE I
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alucent Biomedical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1061-002
Record Dates: First submitted 2022-07-08; First posted 2022-07-13 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: PAD - Peripheral Arterial Disease

STUDY DESIGN:
Intervention Model Description: This study is a prospective, nonrandomized, multicenter, open-label feasibility study of the VRS for the treatment of atherosclerotic de novo or restenotic lesions in the SFA and/or PA after sub-optimal PTA or atherectomy angiographic outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Combination Product: Vessel Restoration System (VRS) — The VRS includes the following components:
  * VRS 10-8-10 Dimer Coated Balloon Catheter
  * VRS Light Fiber
  * VRS Light Source The VRS will collectively refer to all the components used to perform the procedure. Their specific product name will identify individual elements.

SUMMARY:
Feasibility Study of the Vessel Restoration System (VRS) for the Treatment of Atherosclerotic Lesions in the Superficial Femoral Artery (SFA) and/or Popliteal Artery (PA) after Sub-optimal percutaneous transluminal angioplasty (PTA) or Atherectomy: REACTIVATE I

ELIGIBILITY:
Inclusion Criteria:

Subjects for this study must meet all of the following general eligibility criteria

AND the answer must be "YES" to all general inclusion criteria:

1. Subject (or Legal Guardian) is willing and able to provide consent before any study-specific tests or procedures are performed and agree to attend all required follow-up visits.
2. Male or female subject of at least 18 years of age.
3. Chronic symptomatic lower limb ischemia defined as Rutherford classification 2, 3, or 4.
4. Has screen failed from the ACTIVATE II study due to the presence of Grade C or D dissection(s).

Exclusion Criteria:

1. Life expectancy, documented in the Investigator's opinion, of less than 1 year.
2. Cerebrovascular accident (CVA) or transient ischemic attack (TIA) or cardiac event (e.g., PCI for STEMI/NSTEMI, unstable angina) within 6 months prior to the index procedure.
3. Chronic renal insufficiency with serum creatinine ≥ 2.5 mg/dL or eGFR <45 ml/min within 30 days prior to the index procedure or treatment with peritoneal or hemodialysis.
4. Subject has a platelet count < 100,000 cells/mm3 or > 700,000 cells/mm3 within 30 days prior to the index procedure or has a history of bleeding diathesis.
5. Receiving oral or intravenous immunosuppressive therapy.
6. Subject has white blood cell (WBC) count < 3.0 (3,000 cells/mm3) within 30 days prior to the index procedure.
7. History of major amputation in the target limb.
8. Any major intervention planned at the index procedure or within 30 days post-index procedure including treatment of contralateral limb.
9. Subject is pregnant, breastfeeding, or planning to become pregnant in the next 30 days. Subjects (male and female) of childbearing potential must agree to use effective birth control measures for 30 days after the index procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-11-15 (Actual); Primary Completion 2026-11-15 (Estimated); Study Completion 2026-11-15 (Estimated)

PRIMARY OUTCOMES:
An acute reduction in arterial dissections | 12 months
  Reduction in arterial dissection(s) of at least one grade.
Primary Patency as assessed by Doppler Ultrasound (DUS) and freedom from CD-TLR at 1 Year | 12 months
  Primary Patency as assessed by Doppler Ultrasound (DUS)

SECONDARY OUTCOMES:
Technical Success | 12 months
  Technical success is defined by successful delivery of the VRS
Procedural Success | 12 months
  Procedural Success is defined as an acute reduction in arterial dissection(s)
Clinical Success | 36 months
  Clinical success is defined as freedom from CD-TLR
Safety Measure | 72 months
  Frequency of MAEs
Hemodynamic Improvement | 36 months
  Rate of hemodynamic improvement ABI
Rutherford Classification | 36 months
  As assessed by changes in Rutherford Class
Quality of Life Measure | 72 months
  Quality of life (QOL) assessment by EQ-5D

OTHER OUTCOMES:
Major Adverse Limb Events | 36 months
Reintervention for treatment of thrombosis of the target vessel or embolization to its distal Vasculature | 36 months
Major Vascular Complications | 36 months

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - Flinders Medical Center, Adelaide, South Australia
  - The Alfred Hospital, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No
Not sharing IPD